CLINICAL TRIAL: NCT00196053
Title: Observational Registry: The Effectiveness of Pain Management Using the ARCHIMEDES® Implantable Constant-Flow Infusion Pump System for Intrathecal Delivery
Brief Title: The Effectiveness of Pain Management Using the ARCHIMEDES® Constant-Flow Infusion Pump System for Intrathecal Delivery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Codman & Shurtleff (Industry)
Responsible Party: Michael Ward, Worldwide Director, Clinical Research, Codman & Shurtleff
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DDS-EU04-001; EU Pain Registry
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2012-05-02 (Estimated); Status verified 2012-04

CONDITIONS: Chronic Pain
Keywords: Intrathecal pain management; constant flow pump
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Archimedes Constant Flow Implantable Pump

SUMMARY:
The purpose of this observational registry is to collect a continuum of meaningful clinical data on the ARCHIMEDES implantable pump in pain management

DETAILED DESCRIPTION:
Pain management has been a long-standing challenge to the medical community, specifically for the treatment of chronic pain. Chronic Pain is defined by the American Chronic Pain Association as "pain that continues a month or more beyond the usual recovery period for an illness or injury or pain that goes on over months or years as a result of a chronic condition." Chronic pain affects the patient's quality of life, work performance and attendance, mental health, social interactions and overall activities of daily living.

Implantable pumps were used for cancer and non-cancer patients, who had pain, which was resistant to conventional therapy. Intrathecal morphine administration is now accepted as a safe and effective method of controlling or reducing pain and its impact on the sufferer.

The Codman ARCHIMEDES Implantable Constant-Flow Infusion Pump is CE marked, and has been commercially available in Europe for intrathecal delivery of morphine and baclofen since August 1997. ARCHIMEDES is intended for the treatment of chronic intractable (cancer or non-cancer) pain, which requires chronic intrathecal infusion of preservative-free morphine sulfate.

This is a European, multicenter, prospective, single arm, observational registry conducted on a total of 150 Subjects at up to 10 centers in Europe.

Subjects will be followed at 3, 6, 9, and 12 months post Archimedes implant to assess their pain management and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* The Subject has been suffering from chronic (benign and/or malignant) intractable pain for at least 2 or more months duration (pending national laws) with a pre-implant value equal or more than 7 on the Visual Analog Pain Scale.
* The subject does not tolerate oral pain medication at the required therapeutic dose to treat his/her pain.
* The Subject has a minimum reasonable life expectancy of at least 6 months.
* The Subject has given written Informed Consent prior to enrollment into this study.
* The body size of the Subject is sufficient to accept the pump bulk and weight, per the Principal Investigator's discretion.
* The Subject is willing to participate in this registry for 1 year post implant and is willing to comply with the investigational plan requirements.
* It is the Principal Investigator's judgment, based on the knowledge of the Subject, and Subject's condition, as well as the features of the implantable system that the Subject is an appropriate candidate for pain management utilizing an implantable pump for continuously delivering preservative-free morphine sulfate via an intrathecal route.

Exclusion Criteria:

* The Subject has a skin condition (i.e., scleroderma, psoriasis, rash, or open wound) at the site chosen for implantation that would compromise the integrity or access to the injection port.
* The Subject has previously enrolled in or participated in an investigational drug or device trial within the preceding 4 weeks.
* The Subject has any known contraindication to preservative-free morphine sulfate.
* The Subject has a suspected or documented allergy to preservative-free morphine sulfate or related drugs.
* The Subject has a suspected or documented allergy to the materials of the infusion pump or catheter(s) (for example, silicone).
* The Subject has a history of drug and/or alcohol abuse per Principal Investigator discretion.
* The Subject is a female who is pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2005-03; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Pain management measured by the visual analog pain scale | Quarterly for 1 year post-implant
Pain management measured by quality of life score (SF-36) | Quarterly for 1 year post-implant

SECONDARY OUTCOMES:
Device-related adverse events over the duration of the study | End of trial

CONTACTS AND LOCATIONS:
Overall Officials: Michael Ward, DVM, Study Director — Unaffilliated
Locations (8):
- Laon, France
- Germany (5):
  - Bamberg
  - Freiburg im Breisgau
  - Konstanz
  - Meppen
  - Tutzing
- United Kingdom (2):
  - Middlesbrough
  - Plymoth